CLINICAL TRIAL: NCT03865264
Title: Living Organ Donor Recovery Enhancement Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study lost funding
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 015-280
Record Dates: First submitted 2018-02-08; First posted 2019-03-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Living Liver and Kidney Donors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Living Liver donor (Active Comparator): Recovery enhancement program:
  1. At least 6 weeks of physical and relaxation skills training pre-transplant.
  2. Taking nutritional drink for 5 days before and after the surgery.
  3. Opioid sparing pain management.
  Interventions: Other: Recovery Enhancement Program
- Living Kidney donor (Active Comparator): Recovery Enhancement Program
  1. At least 4 weeks of physical and relaxation skills training pre-transplant.
  2. Taking nutritional drink for 5 days before and after the surgery.
  3. Opioid sparing pain management.
  Interventions: Other: Recovery Enhancement Program
- Living Kidney donor (Control) (No Intervention): 1. Subjects maintain the same lifestyle without practicing physical training, relaxation skills or nutritional drink before and after the surgery.
  2. To control post-op pain, subject will use medication per standard of care, including PCA pump.

INTERVENTIONS:
Other: Recovery Enhancement Program — Behavioral, nutritional, physical and opioid-reduction pain medication
  Arms: Living Kidney donor; Living Liver donor

SUMMARY:
The purpose of the study is to test if using these living donor-specific pre-transplant resources would lead to a better and faster recovery post-transplant.

DETAILED DESCRIPTION:
Donor safety and outcomes are the chief concerns of programs performing living donor liver and kidney transplantation. The protection of donors from physical and emotional harm has been a fundamental principle in living donor liver and kidney donation from the beginning. The safety of living donor hepatectomy and nephrectomy has been established. The risks associated with the donation have been deemed acceptable by the transplant community.

The investigators would like to move beyond the safety of the operation and address the most important post-operative issues that potentially cause donors physical and emotional stress: these include pain control, appropriate nutrition for optimal liver regeneration and physical/functional recovery, fatigue, time to return to normal physical and work activity, and difficulties coping with recovery and any possible complications. The goal of conducting this study is to create a program of pre- and post-operative interventions to enhance recovery so that patients can return to their normal quality of life as soon as possible. Currently there is no literature on programs to enhance living donor care and recovery.

This study will be conducted to determine if interventions during the pre-operative (a minimum of four weeks in an exercise program), intra-operative (anesthesia), and post-operative (pain management) stages have an effect on liver and kidney donor patients' quality of life and return to baseline functional status.

ELIGIBILITY:
Inclusion Criteria:

1. Ages ≥ 18 years
2. Cleared by a physician to participate in an exercise program
3. Approved for evaluation to be a living liver or kidney donor
4. Subjects willing and able to comply with the protocol procedures for the duration of the study, including the exercise regimen and scheduled follow-up visits
5. Subjects who have given IRB-approved written informed consent, prior to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care

Exclusion Criteria:

1. Any co-morbidity restricting the subject's ability to walk alone
2. Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
RAND SF-36 questionnaires | From day of enrollment in the study (at least 4 weeks before surgery) up to 1 day prior to hepatectomy.
  Pre-operative emotional stress
Level of pain experienced daily | From day of admission into ICU (post-hepatectomy) up to day of hospital discharge (4-14 days post-hepatectomy)
  level of pain per numerical rating pain scale (scale 0-10) with 0 being no pain and 10 being severe pain.
Duration in ICU | From day admission into ICU up to day of discharge to hospital floor or 14 days post hepatectomy, whichever came first.
  Duration in ICU post-hepatectomy
Opioid usage | From day of hospital discharge (post-hepatectomy) up to 1 year post hepatectomy.
  Number of participants that require using opioid medication to treat abdominal and incisional pain post hepatectomy, medication strength and frequency of use.
RAND SF-36 questionnaires | From month 1 to month 12 post transplantation.
  Post-operative emotional stress
Duration to return of daily activities | From day of hospital discharge to 1 year follow up.
  Duration to return of daily activities
Incidence of Post-operative hospital re-admissions | From post-transplant discharge to 1 year follow-up
  Number of post-operative hospital re-admissions

CONTACTS AND LOCATIONS:
Overall Officials: Guiliano Testa, MD, Principal Investigator — Simmons Transplant Institute, Baylor University Medical Center
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States